CLINICAL TRIAL: NCT06161662
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Postoperative Delirium and EEG Characteristic Parameters in Elderly Patients Undergoing Abdominal Surgery Under General Anesthesia
Brief Title: Effect of Acupoint Stimulation on Postoperative Delirium and Electroencephalogram
Acronym: AS-DEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XJH-A-20230920
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia; Postoperative Delirium; Electroencephalogram
Keywords: Transcutaneous electrical acupoint stimulation; Postoperative delirium; Electroencephalogram
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Four or six patients were defined as a block group and the results were sealed in envelopes using computer-generated block randomisation by a researcher not involved in clinical anesthesia. After the patients were enrolled, the study nurse opened the envelope according to the corresponding enrollment number and obtained the group results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical stimulation (Experimental): At the beginning of anesthesia induction, the electrodes are attached to the skin at the Neiguan point and Shenmen point and connected to the percutaneous acupoint electrical stimulation device (Hwato , Suzhou Medical Equipment Factory). Electrical stimulation is given.
  Interventions: Other: transcutaneous electrical acupoint stimulation
- Control (Other): At the beginning of anesthesia induction, the electrodes are attached to the skin at the Neiguan point and the Shenmen point without stimulation
  Interventions: Other: Control

INTERVENTIONS:
Other: transcutaneous electrical acupoint stimulation — Electrodes will be attached on the surface of acupoints and electrical stimulation will be given
  Other Names: TEAS
  Arms: Transcutaneous electrical stimulation
Other: Control — Electrodes will be attached on the surface of acupoints but no stimulation will be given
  Arms: Control

SUMMARY:
Transcutaneous electrical acupoint stimulation (TEAS) was reported to benefit the patients undergoing surgeries by reducing anesthetics consumption and decreasing anesthesia related adverse effects. Electroencephalogram (EEG) and EEG-related indicators are important indicators reflecting the conscious state of the brain, and different anesthetic drugs and anesthesia depths cause different EEG characteristic changes. The mechanism by which TEAS improves postoperative delirium (POD) is not clear, and whether changes in EEG characteristic parameters is involved needs to be further explored. Therefore, this study aims to observe the effect of TEAS at Neiguan and Shenmen acupoint on POD in elderly patients undergoing abdominal surgery, and to explore the EEG related mechanism underlying TEAS improving POD.

ELIGIBILITY:
Inclusion Criteria:

1. aged 65 years or older
2. American Society of Anesthesiologists (ASA) classification≤ Grade III
3. Patients scheduled for elective abdominal surgery under general anesthesia
4. Informed consent

Exclusion Criteria:

1. Patients with severe central nervous system injury or severe cerebrovascular disease
2. Patients with cognitive dysfunction assessed by Confusion Assessment Method before surgery
3. Patients unable to cooperate with studies, such as psychiatric disorders or difficulty in communication
4. Patients with severe hepatic and renal insufficiency
5. Patients with severe respiratory diseases
6. Patients with contraindication for transcutaneous electrical stimulation, such as implanted electrophysiological devices, skin infection and damage at acupuncture points
7. Anticipated duration of anesthesia shorter than 2 hours or postoperative hospital stay shorter than 3 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium by 7 days after surgery | from end of surgery to 7 days after surgery
  Delirium will be assessed by 3-minute Diagnostic Interview for Confusion Assessment Method

SECONDARY OUTCOMES:
maximal electroencephalogram (EEG) alpha band power reduction | From anesthesia induction to the end of surgery
Maximal decrease of regional cerebral oxygen saturation | From anesthesia induction to the end of surgery
EEG explosive suppression time | From anesthesia induction to the end of surgery
  EEG burst suppression is defined as a burst-suppression ratio (BSR) ≥ 10%, more than 1 minute
Incidence of major neurological complications | From end of surgery to discharge from hospital, at an average of 7 days
  Coma, stroke, altered state of consciousness
The Athens Insomnia Scale and Epworth somnolence Scale score by 1 day after surgery | From end of surgery to 1 day after surgery
The Athens Insomnia Scale and Epworth somnolence Scale score by 3 days after surgery | From end of surgery to 3 days after surgery
The Hospital Anxiety and Depression Scales by 1 day after surgery | From end of surgery to 1 day after surgery
The Hospital Anxiety and Depression Scales by 3 days after surgery | From end of surgery to 3 days after surgery
The Quality of Recovery-15 Score by 1 day after surgery | From end of surgery to 1 day after surgery
The Quality of Recovery-15 Score by 3 days after surgery | From end of surgery to 1 day after surgery
Incidence of delirium by 1 day after surgery | From end of surgery to 1 day after surgery
Incidence of delirium by 3 days after surgery | From end of surgery to 3 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of the Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
individual data including protocol and statistical analysis plan will be shared during 3 months and 5 years following article publication after deidentification
Supporting Information: SAP
Time Frame: during 3 months and 5 years following article publication after deidentification

REFERENCES:
- [Background] Guay CS, Kafashan M, Huels ER, Jiang Y, Beyoglu B, Spencer JW, Geczi K, Apakama G, Ju YS, Wildes TS, Avidan MS, Palanca BJA. Postoperative Delirium Severity and Recovery Correlate With Electroencephalogram Spectral Features. Anesth Analg. 2023 Jan 1;136(1):140-151. doi: 10.1213/ANE.0000000000006075. Epub 2022 May 13. PMID 36130079
- [Background] Feng B, Zhang Y, Luo LY, Wu JY, Yang SJ, Zhang N, Tan QR, Wang HN, Ge N, Ning F, Zheng ZL, Zhu RM, Qian MC, Chen ZY, Zhang ZJ. Transcutaneous electrical acupoint stimulation for post-traumatic stress disorder: Assessor-blinded, randomized controlled study. Psychiatry Clin Neurosci. 2019 Apr;73(4):179-186. doi: 10.1111/pcn.12810. Epub 2019 Jan 22. PMID 30565342

DOCUMENTS (2):
  • Study Protocol (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT06161662/Prot_000.pdf
  • Informed Consent Form (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT06161662/ICF_001.pdf